CLINICAL TRIAL: NCT04173624
Title: Endosonography Versus Magnetic Resonance Cholangiopancreatography for Choledocholithiasis for Intermediate Risk of Choledocholithiasis (as Per European Society of Gastrointestinal Endoscopy Guidelines )- Randomized Controlled Trial
Brief Title: To Compare EUS and MRCP in Detecting Choledocholithiasis in Patients of Intermediate Risk of Choledocholithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh K, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EUS Vs MRCP-01
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Choledocholithiasis
Keywords: EUS; MRCP; Intermediate Probability
MeSH Terms: conditions — Choledocholithiasis | interventions — Endosonography; Cholangiopancreatography, Magnetic Resonance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endosonography (Experimental): Endosonography is endoscopic method to diagnose pancreatic and biliary disorders. Participants randomized to this arm will undergo diagnostic endosonography under propofol sedation in supervision of trained anesthesiologists. If choledocholithiasis is diagnosed on endosonography, patient will be subjected for endoscopic retrograde cholangiopancreatography for clearance of stone. If choledocholithiasis is not present then participants will be kept in follow-up and further evaluation will be done if clinically indicated as per discretion of treating physician.
  Interventions: Diagnostic Test: Endosonography
- Magnetic Resonance Cholangiopancreatography (Experimental): Magnetic Resonance Cholangiopancreatography (MRCP) is non-invasive method for diagnosis of pancreatic and biliary disorders. Participants randomized to this arm will undergo MRCP. If choledocholithiasis is diagnosed on MRCP, participants will be subjected for endoscopic retrograde cholangiopancreatography for clearance of stone. If choledocholithiasis is not present then participants will be kept in follow-up and further evaluation will be done if clinically indicated as per discretion of treating physician.
  Interventions: Diagnostic Test: Magnetic Resonance Cholangiopancreatography

INTERVENTIONS:
Diagnostic Test: Endosonography — Endosonography (EUS) is endoscopic method for evaluated pancreatic and biliary pathology.
  Arms: Endosonography
Diagnostic Test: Magnetic Resonance Cholangiopancreatography — Magnetic Resonance Cholangiopancreatography (MRCP) is non-invasive method for evaluating pancreatic and biliary pathology
  Arms: Magnetic Resonance Cholangiopancreatography

SUMMARY:
A Recent Meta analysis, showed pooled sensitivity and specificity were 97% and 90 for EUS and 87% and 92 for MRCP . This meta analysis includes only 5 studies, smaller sample size in each study, significant heterogeneity in reference standards ranged from ERCP and Intra operative cholangiography (IOC) to clinical follow up for negative patients . Furthur validation of EUS Vs MRCP is needed in detecting common bile duct caliculi in intermediate risk of choledocholithiasis To date Randamized control trail comparing EUS Vs MRCP in detecting Choledocholithiasis lacking , hence the investigators aimed a Randamized control trail determining and comparing the sensitivity and specificity of EUS and MRCP in diagnosing Choledocholithiasis.

DETAILED DESCRIPTION:
Aim: Endosonography Versus Magnetic Resonance Cholangiopancreatography for Choledocholithiasis for Intermediate Risk of Choledocholithiasis (as Per European Society of Gastrointestinal Endoscopy Guidelines )- Randomized Controlled Trial

Outcomes

A.Primary Outcome :

•Sensitivity and Specificity of EUS Vs MRCP

B.Secondary Outcomes:

* Cost effectiveness
* Adverse effects
* Additional Clinically Significant endoscopic findings

MATERIAL AND METHODS Study area •out-patients and in-patients in Asian Institute of Gastroenterology Study design Randamized control study Study period November 2019-March 2020

INCLUSION CRITERIA:

•Patients over 18yrs of age with suspected choledocholithiasis stratified into intermediate risk of choledocholithiasis as per European Society of Gastrointestinal Endoscopy Guidelines Guidelines

Exclusion criteria:

* Patients with Cholangitis
* Patients with hypotension
* Ultrasound or CT cross sectional image showing stone
* Patients with contraindications to MRCP (claustrophobia ,pacemaker, or any prosthesis contraindicating MR)
* Predictable impossibility to perform a complete exploration of pancreato biliary area by EUS (gastroenteroanastomosis or stenosis )
* Patients with suspected pancreato biliary malignancy or pancreato biliary malformations
* Patients with history significant alcohol intake
* Patients taking hepato toxic drugs
* Patients in whom serum hepatitis B or C antibodies are present
* Patients with confirmed history of choledocholithiasis or history of biliary sphincterotomy
* Patients not giving consent for participation

STUDY PROCEDURE The study will be a Randomized control study where sensitivity and specificity and secondary outcomes - cost effectiveness, adverse effects will be compared between EUS and MRCP group . All the patients presented to outpatient department or in patient wards with suspected choledocholithiasis will be screened as per European Society of Gastrointestinal Endoscopy guideline. Patients stratified into intermediate probability will be selected based on inclusion and exclusion criteria. Then patients will randomized to either EUS or MRCP based computerized software .Patients who are randomized to EUS group will undergo EUS for detection of Choledocholithiasis and then undergo Endoscopic Retrograde Cholangiopancreatography (ERCP) at same time if calculi detected and patients in whom calculi was not found, management is based on clinical judgement and 3months follow up . Patients who are randomized to MRCP group will undergo MRCP for detection of Choledocholithiasis and then undergo ERCP if calculi detected. Patients in whom calculi was not found, management will be based on clinical judgement and 3 months follow up. Based on presence of or absence of stone in Reference standard i.e in ERCP following EUS or MRCP or during 3 month follow up , sensitivities and specificities of EUS and MRCP are calculated and compared .

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18yrs of age with suspected choledocholithiasis stratified into intermediate risk of choledocholithiasis as per European Society of Gastrointestinal Endoscopy Guidelines

Exclusion Criteria:

* Patients with Cholangitis
* Patients with hypotension
* Ultrasound or CT cross sectional image showing stone
* Patients with contraindications to MRCP (claustrophobia ,pacemaker, or any prosthesis contraindicating MR)
* Predictable impossibility to perform a complete exploration of pancreato biliary area by EUS (gastroenteroanastomosis or stenosis )
* Patients with suspected pancreato biliary malignancy or pancreato biliary malformations
* Patients with history significant alcohol intake
* Patients taking hepato toxic drugs
* Patients in whom serum hepatitis B or C antibodies are present
* Patients with confirmed history of choledocholithiasis or history of biliary sphincterotomy
* Patients not giving consent for participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of EUS Vs MRCP | 4 month
  This study will evaluate diagnostic accuracy of MRCP and EUS in patients with intermediate probability of choledocholithiasis as per European society of GI endoscopy guidelines

SECONDARY OUTCOMES:
Rate of Adverse Events | 4 month
  Adverse events related with EUS and MRCP will be collected. Those who undergo ERCP for choledocholithiasis, total adverse events related to ERCP will be collected.
Cost - Effectiveness | 4 months
  Cost benefits analysis for EUS Vs MRCP will be done for detection of choledocholithiasis by using total cost along with direct and indirect cost.
Rate of Additional Significant Endoscopic finding | 4 months
  In Endosonography arm, total additional endoscopic clinically significant findings such as ulcer, polyps, esophageal and gastric varies, gastric outlet obstruction will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

REFERENCES:
- [Derived] Jagtap N, Kumar JK, Chavan R, Basha J, Tandan M, Lakhtakia S, Kalapala R, Nabi Z, Gupta R, Ramchandani M, Talukdar R, Reddy M, Yarlagadda R, Singh J, Memon SF, Venkat Rao G, Reddy DN. EUS versus MRCP to perform ERCP in patients with intermediate likelihood of choledocholithiasis: a randomised controlled trial. Gut. 2022 Feb 10:gutjnl-2021-325080. doi: 10.1136/gutjnl-2021-325080. Online ahead of print. PMID 35144973